CLINICAL TRIAL: NCT04210869
Title: The Long-Term Effects of Mixed Nuts Consumption on Brain Vascular Function in Elderly Men and Women
Brief Title: Mixed Nuts and Brain Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: The International Nut and Dried Fruit Council (INC) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: METC 19-058
Record Dates: First submitted 2019-12-18; First posted 2019-12-26 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Brain Vascular Function; Cerebral Blood Flow
Keywords: Brain Insulin Sensitivity; Cognitive Performance

STUDY DESIGN:
Intervention Model Description: Crossover Assignment Participants will receive, in random order, daily 60 g of mixed nuts (mixed nut treatment) or no food products (control treatment) for sixteen weeks, separated by a washout period of at least 8 weeks.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Mixed nuts
  Interventions: Dietary Supplement: Mixed Nuts
- Control (No Intervention): No mixed nuts

INTERVENTIONS:
Dietary Supplement: Mixed Nuts — Study volunteers will receive daily 60 g of mixed nuts (15 g walnut, 15 g cashew, 15 g hazelnut, 15 g pistachio) for 16 weeks.
  Arms: Experimental

SUMMARY:
Impaired brain vascular function precedes the development of reduced cognitive performance, while brain insulin-resistance is also associated with cognitive decline. The Mediterranean diet, which is rich in nuts, may protect against the development of impaired cognitive performance. The hypothesis is that long-term mixed nut consumption increases brain insulin-sensitivity thereby improving brain vascular function and cognitive performance. The primary objective is to evaluate in elderly men and women the effect of 16-week mixed nut consumption on cerebral blood flow, as quantified by the non-invasive gold standard magnetic resonance imaging (MRI)-perfusion method Arterial Spin Labelling (ASL). Cerebral blood flow is a robust and sensitive physiological marker of brain vascular function. Secondary objectives are to investigate effects on the cerebral blood flow response to intranasal insulin delivery - a marker of insulin-sensitivity in the human brain - as quantified by ASL, and cognitive functioning as assessed with a neuropsychological test battery.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 60-70 years
* BMI between 25-35 kg/m2
* Fasting plasma glucose < 7.0 mmol/L
* Fasting serum total cholesterol < 8.0 mmol/L
* Fasting serum triacylglycerol < 4.5 mmol/L
* Systolic blood pressure < 160 mmHg and diastolic blood pressure < 100 mmHg
* Stable body weight (weight gain or loss < 3 kg in the past three months)
* Willingness to give up being a blood donor from 8 weeks before the start of the study, during the study and for 4 weeks after completion of the study
* No difficult venipuncture as evidenced during the screening visit

Exclusion Criteria:

* Allergy or intolerance to nuts
* Left-handedness
* Current smoker, or smoking cessation < 12 months
* Diabetic patients
* Familial hypercholesterolemia
* Abuse of drugs
* More than 3 alcoholic consumptions per day
* Use of products or dietary supplements known to interfere with the main outcomes as judged by the principal investigators
* Use medication to treat blood pressure, lipid or glucose metabolism
* Use of an investigational product within another biomedical intervention trial within the previous 1-month
* Severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* Active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident
* Contra-indications for MRI imaging (e.g. pacemaker, surgical clips/material in body, metal splinter in eye, claustrophobia)

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Brain Vascular Function | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Cerebral blood flow as quantified non-invasively by the MRI perfusion method Arterial Spin Labeling (ASL)

SECONDARY OUTCOMES:
Brain Insulin Sensitivity | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Change in cerebral blood flow, as quantified non-invasively by the MRI perfusion method Arterial Spin Labeling (ASL), before and after application of intranasal insulin (160 IU)
Cognitive performance | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Cambridge Neuropsychological Test Automated Battery (CANTAB)

OTHER OUTCOMES:
Glucose metabolism | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Oral Glucose Tolerance Test (OGTT)
Peripheral vascular function (1) | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Flow-mediated vasodilation (FMD)
Peripheral vascular function (2) | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Carotid artery reactivity (CAR)
Peripheral vascular function (3) | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Pulse wave analysis (PWA)
Peripheral vascular function (4) | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Pulse wave velocity (PWV)
Peripheral vascular function (5) | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Retinal microvascular calibers
Blood pressure | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Office and 24-hour ambulatory blood pressure
Advanced glycation endproducts | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Serum protein-bound advanced glycation endproducts (AGEs)
Blood lipids | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Lipids and Lipoproteins
Blood glucose | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Glucose
Blood insulin | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Insulin
Blood markers for low-grade systemic inflammation | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Markers for low-grade systemic inflammation (IL-6, TNF-alpha)
Blood markers for microvascular function | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Markers for microvascular function (sCAM-1, vWf, cGMP)
Blood marker of neurogenesis | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Brain-derived neurotrophic factor
Parameters for compliance | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Alpha-linoleic acid levels (blood)
Structural brain status | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  MRI Structural MPRAGE scan
Functional connectivity | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Resting and task-induced blood-oxygen-level-dependent (BOLD) response, as quantified by functional MRI T2*-weighted imaging.
Fat distribution in abdomen | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Magnetic Resonance Imaging measurements will be included to quantify abdominal fat compartments (i.e.
  subcutaneous and visceral fat) and fat content of abdominal organs (i.e. liver and pancreas).
Microbiota composition | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Fecal samples will be collected to be used for analysing different species of microbiota.
Other perceivable benefits: Quality of Life | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  The Quality of life will be assessed using a 32-item questionnaire
Other perceivable benefits: Sleep characteristics | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Sleep characteristics will be assessed using the 10-item Pittsburgh Sleep Quality Index
Other perceivable benefits: Mood | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Mood will be tested using the Affect Grid
Other perceivable benefits: Physical fitness (1) | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Timed up-and-go test (TUGT)
Other perceivable benefits: Physical fitness (2) | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  The 6-minute walk test (6 MWT)
Other perceivable benefits: Physical fitness (3) | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Handgrip test
Other perceivable benefits: Physical fitness (4) | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Muscle strength test, as measured using the Biodex system
Weight | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Weight in kilograms
Length | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Length in meters
Waist circumference | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Waist circumference in centimeters
Hip circumference | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Hip circumference in centimeters
Indirect fat distribution | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Measured by skinfold measurements
Food intake | Change in outcomes at the end of a 16-week mixed nuts intervention and 16-week control period.
  Food intake will be assessed using the Food Frequency Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Joris, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Nijssen KM, Mensink RP, Plat J, Ivanov D, Preissl H, Joris PJ. Mixed nut consumption improves brain insulin sensitivity: a randomized, single-blinded, controlled, crossover trial in older adults with overweight or obesity. Am J Clin Nutr. 2024 Feb;119(2):314-323. doi: 10.1016/j.ajcnut.2023.12.010. Epub 2023 Dec 20. PMID 38128733